CLINICAL TRIAL: NCT01904240
Title: Lipopolysaccharide Binding Protein as a Potential Biomarker of Parkinson's Disease
Brief Title: Evaluation of a Biomarker Related to the GI Tract for the Diagnosis of Parkinson's Disease
Status: Completed | Type: Observational
Sponsor: Rush University Medical Center (Other)
Responsible Party: Sponsor
Other Study IDs: 12102401-IRB01
Record Dates: First submitted 2013-07-09; First posted 2013-07-22 (Estimated); Last update posted 2014-11-13 (Estimated); Status verified 2014-11

CONDITIONS: Parkinson's Disease
Keywords: Parkinson's disease; GI tract; Lipopolysaccharide binding protein
MeSH Terms: conditions — Parkinson Disease

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Cross-Sectional
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (2):
- Parkinson's disease patients: Patients with Parkinson's disease
- Subjects without Parkinson's disease: Control subjects without Parkinson's disease

SUMMARY:
The cause of Parkinson's disease (PD) is currently unknown. Both environmental and genetic factors have been found to contribute to PD pathogenesis. The pathology of PD is distributed throughout the entire nervous system including the central, peripheral, and enteric nervous system. There is evidence that inflammation plays a major role in neurodegeneration in PD. In both the striatum and substantia nigra of PD patients activated microglia were found and proinflammatory cytokines (TNF, IL-1B, IL-6, iNOS) are increased in the CSF. An inflammation-driven animal model has emerged and has been widely accepted as a model of the disease based on lipopolysaccharide (LPS) induced neurotoxicity. LPS is an endotoxin found on the outer membrane of gram negative bacteria and humans are exposed to LPS through the intestinal tract. The intestinal tract and thus the enteric nervous system serve as a conduit to the central nervous system. It has been posited that the inflammatory process could gain access to the lower brainstem via the vagal nerve and then ascend through the basal mid- and forebrain until it reaches the cerebral cortex, producing various pre-motor and motor symptoms of PD along the way. LPS may be one of the inflammatory triggers involved in this process. Systemic exposure to bacterial endotoxin can be determined by measuring plasma LPS binding protein (LBP). A study of 9 patients with early PD (median Hoehn and Yahr stage 2) and age matched controls found that the PD subjects had a significantly lower mean level of plasma LBP compared to control subjects. The aim of the research plan is to establish LBP as a potential biomarker for PD across a spectrum of disease severity.

ELIGIBILITY:
Inclusion Criteria for Parkinson's disease subjects:

* Patients with a clinical diagnosis of Parkinson's disease by United Kingdom Parkinson Disease Society Brain Bank criteria will be recruited.
* Hoehn and Yahr stage 1-5
* Parkinson's disease symptomatic treatment will be allowed.

Exclusion Criteria for Parkinson's disease subjects:

* Treatment with medications that may induce parkinsonism (metoclopramide, typical, or atypical antipsychotic agents)
* Known diagnosis of inflammatory bowel disease.
* Symptomatic functional GI disease that significantly impairs intestinal mobility such as scleroderma or use of GI motility drugs.
* Acute illness requiring immediate hospitalization.
* Presence of short bowel syndrome or severe malnutrition with ideal body weight < or = 90%

Inclusion Criteria for control subjects:

* No evidence of GI symptoms other than minor hematochezia attributable to hemorrhoids.
* No evidence of symptoms of Parkinson's disease.
* Matching in age and gender to the Parkinson's disease patients.

Exclusion Criteria for control subjects:

* Presence of Parkinson's disease or its symptoms.
* Treatment with medications that may induce parkinsonism (metoclopramide, typical, or atypical antipsychotic agents)
* Known diagnosis of inflammatory bowel disease.
* Symptomatic functional GI disease that significantly impairs intestinal mobility such as scleroderma or use of GI motility drugs.
* Acute illness requiring immediate hospitalization.
* Presence of short bowel syndrome or severe malnutrition with ideal body weight < or = 90%

Ages: 30 Years to 90 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: Rush University Movement Disorders Clinic
Sampling Method: Non-Probability Sample
Enrollment: 200 (Actual)
Dates: Start 2013-07; Primary Completion 2014-06 (Actual); Study Completion 2014-06 (Actual)

PRIMARY OUTCOMES:
Lipopolysaccharide binding protein (LBP) level | one day
  measure serum and plasma LBP levels in PD patients and control subjects

CONTACTS AND LOCATIONS:
Overall Officials: Gian D Pal, MD, Principal Investigator — Rush University Medical Center
Locations (1):
- Rush University Medical Center, Chicago, Illinois, United States